CLINICAL TRIAL: NCT00571051
Title: MEG Study of Mindfulness Based Stress Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Kerr, Catherine, Associate Professor, Harvard Medical School (HMS and HSDM)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: K01AT003459 (NIH); 001
Record Dates: First submitted 2007-12-07; First posted 2007-12-11 (Estimated); Last update posted 2019-09-11 (Actual); Status verified 2009-08

CONDITIONS: Somatosensory Cortical Dynamics in Normal Humans
Keywords: MEG, mindfulness, tactile perception
MeSH Terms: interventions — Mindfulness-Based Stress Reduction; Mindfulness

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- 1 (Experimental): MBSR 8 week course
  Interventions: Behavioral: Mindfulness Based Stress Reduction
- 2 (No Intervention): 8 weeks of natural history

INTERVENTIONS:
Behavioral: Mindfulness Based Stress Reduction — 8 week course in mindfulness training
  Other Names: Course is modelled on course taught by Center for Mindfulness, UMASS Worcester. Instructor and lesson plan are certified by Center for Mindfulness
  Arms: 1

SUMMARY:
The purpose of this research is to investigate the effects of mindfulness based stress reduction (MBSR) on measures of brain function. We are looking especially at the ways in which MBSR may affect the way the brain processes the sense of touch. The study seeks to recruit healthy, normal adults who are interested in MBSR training, a simple program that involves learning how to pay attention mindfully to the present moment

DETAILED DESCRIPTION:
In this study, investigators will randomly assign volunteers to one of two conditions: (1) attend classes to learn MBSR (2) be on a waitlist on which volunteers will continue your activities until the conclusion of the study, at which point they will be offered free MBSR training. The MBSR class and the body scan classes will be videotape-recorded in order to ensure that the instruction meets study standards. Since the videotape will capture your image and voice, you will be identifiable. However, this videotape will only be viewed by HIPAA certified study staff; it will be stored in a locked drawer and will be destroyed 36 months after the completion of the study.

Random assignment works like the flip of a coin. A volunteer has a 1 in 3 chance of receiving MBSR, being asked to continue with his or her normal life, or being asked to practice body scanning. At any time and for any reason at all a volunteer may decide to withdraw from the study. Data about volunteers' experiences, brain structure, and function collected from this study will be stored by investigators at the Osher Institute, Harvard Medical School.

If a volunteer is randomly assigned to receive MBSR, he or she will be asked to attend 8 class sessions of training which will last 2 hours each. He or she will also be asked to attend a 5 hour retreat. In MBSR classes, you will receive instruction in mindfulness based body scan meditation. In addition, a subject assigned to MBSR will receive instruction in sitting meditation and in gentle yoga. Participants in both classes will also be asked to reflect on their meditation experiences during class and will be asked to consider carrying out a home practice during the week, outside of class. MBSR and body scan classes will meet at a meditation class facility convenient to a red line T stop in Cambridge.

Study assessment visits to the Martinos Center facility in Charlestown

In this study, there are 3 study assessment visits to the Martinos Center facility in Charlestown in which volunteers will be asked questions about their daily experience. At all 3 study visits, investigators will also record magnetic field readings of the brain using a non-invasive imaging technique known as magnetoencephalography (MEG). MEG is a technique that measures the small electrical currents produced when cells in the brain are active. This activity is sometimes called "brain waves."

During these recordings, we will also be lightly touching volunteers' left hand and left foot with a plastic knob. We will be asking volunteers to tell us when they think that they can the stimulus.

To help us interpret the MEG magnetic field readings, at a volunteer's first visit we will also use magnetic resonance imaging (MRI) to create an image of his/her brain. MRI is a technique that uses magnetic fields to align the spinning of atoms in water molecules. It then creates an image of the brain and its activity from the tiny amounts of energy released when the atoms relax to their normal state. Structural MRI will give us information about the anatomy of the brain.

At each of the 3 study visits, before a subject begins the brain scans, he/she will be asked to complete two tests. The first test has an assistant lightly press plastic domes on his/her fingertips. The domes have grooves, and he/she will be asked to tell us which way the grooves point. The second test asks him/her to find numbers that will appear on a screen with flashing letters.

Volunteers will also be given questions about daily experience. In addition, at visits 2 and 3, if a subject is assigned to receive MBSR, investigators will ask about experiences with MBSR practice.

Schedule of assessment procedures in visits 1-3:

* Visit 1 involves the following procedures:

  * Receiving a magnetic resonance imaging (MRI) brain scan.
  * Doing the dome test and numbers test
  * Filling out brief questionnaires about activities that performed with the hand, and feelings and experiences in general.
  * Undergoing a magnetoencephalography (MEG) recording of brain function.
* Visit 2 involves the following procedures:

  * Doing the dome test and numbers test
  * Filling out brief questionnaires about feelings and experiences in general and feelings and experiences related to MBSR.
  * Undergoing a magnetoencephalography (MEG) recording of brain function.
* Visit 3 involves the following procedures:

  * Doing the dome test and numbers test
  * Filling out brief questionnaires about feelings and experiences in general and feelings and experiences related to MBSR.
  * Undergoing a magnetoencephalography (MEG) recording of brain function.

Each of the 3 study visits to the Martinos Center will last up to 2 hours and 30 minutes.

Optional MBSR class for subjects assigned to waitlist

If a subject is assigned to the waitlist, he/she will have the option of enrolling in a free MBSR class after the completion of study visits to the Martinos Center. This free class will be taught by the chief mindfulness teacher who is a certified MBSR instructor. This free class is offered to only as a courtesy expression of thanks for participating in this study. This free class is not a research study: no research data will be collected in this courtesy class; subjects are free to participate or to refuse to participate in this post-study optional class.

ELIGIBILITY:
Inclusion Criteria:

-

You are eligible to participate in this study because you meet all of our selection criteria:

* You are between ages 18-50
* You are right-handed
* You are able to receive a MRI scan (you have no metal implants or other metal objects or medical devices that would make a MRI scan unsafe for you)
* You are able to follow study instructions and can read and write English

Exclusion Criteria:

* You are not eligible to participate in this study if you:

  * have any systemic musculoskeletal diseases such as rheumatoid arthritis, systemic lupus, or scleroderma that would affect the function of your nervous system
  * have any neurological conditions that might affect your hand, wrist, or arm function
  * respond to our questionnaires in a manner suggesting you may be suffering from depression
  * are pregnant or a nursing mother
  * currently have any ongoing meditation practice, including MBSR.
  * are unable to complete our study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-10; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Somatosensory cortical dynamics | 8 weeks

SECONDARY OUTCOMES:
Rumination; mindfulness; somatosensory evoked potentials; tactile thresholds | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Kerr, PhD, Principal Investigator — Harvard Medical School (HMS and HSDM)
Locations (1):
- Harvard Medical School, Boston, Massachusetts, United States

REFERENCES:
- [Background] Kerr CE, Wasserman RH, Moore CI. Cortical dynamics as a therapeutic mechanism for touch healing. J Altern Complement Med. 2007 Jan-Feb;13(1):59-66. doi: 10.1089/acm.2006.5245. PMID 17309379